CLINICAL TRIAL: NCT01291901
Title: A Phase II, Randomized, Double Blind, Placebo-controlled, Multicenter Study to Investigate the Impact of NP2 in Subjects With Intractable Pain Due to Malignancy
Brief Title: NP2 Enkephalin For Treatment of Intractable Cancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diamyd Inc (Industry)
Collaborators: Paragon Biomedical (Industry); invivodata, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP2/P2/10/2
Record Dates: First submitted 2011-02-04; First posted 2011-02-09 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Intractable Pain; Neoplasms
Keywords: pain; cancer; malignancy; intractable; gene therapy; enkephalin; opioid
MeSH Terms: conditions — Pain, Intractable; Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active NP2 (Experimental): Single intradermal dose of active NP2. An open label study extension will offer up to two additional doses of active NP2 between weeks 4-10 following the previous dose.
  Interventions: Biological: NP2
- Placebo (Placebo Comparator): Single intradermal dose of placebo (vehicle). An open label study extension will offer up to two additional doses of active NP2 between weeks 4-10 following the previous dose.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NP2 — NP2 is a replication defective HSV-1 based gene transfer vector engineered to express human preproenkephalin. The drug will be injected intradermally corresponding to the distribution of the malignancy-related pain. The total amount to be injected will be a dose volume of 1.0 ml delivered in a single session on Study Day 0.
  Arms: Active NP2
Biological: Placebo — The placebo (vehicle) will be injected intradermally corresponding to the distribution of the malignancy-related pain. The total amount to be injected will be a dose volume of 1.0 ml delivered in a single session on Study Day 0.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the impact of intradermal delivery of NP2 on pain scores and pain medication usage in subjects with intractable pain due to malignant disease. A second purpose is to confirm safety and secondary efficacy measurements.

DETAILED DESCRIPTION:
Chronic severe pain remains a significant unmet medical need in patients that have progressive cancer. Existing treatments have limited efficacy and also suffer significant side effects. This is a multi-center, randomized, double blind, placebo-controlled clinical trial designed to evaluate the impact of intradermal injection of NP2 in subjects who have intractable pain due to malignant disease. NP2 is a gene transfer vector engineered to express human preproenkephalin, a gene naturally involved in pain control. Delivery of NP2 directly to the site of pain caused by cancer is intended to provide increased Enkephalin peptides, which bind to opioid receptors, that may allow better pain control.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed malignant disease.
* Intractable pain related to malignancy.
* Females must be postmenopausal or practicing birth control.
* Able to provide appropriate written consent.

Main Exclusion Criteria:

* Positive pregnancy test prior to receiving study treatment.
* Serious uncontrolled medical condition other than malignancy (e.g. congestive heart failure, coagulopathy, uncontrolled diabetes).
* Evidence of active Hepatitis B, Hepatitis C, or HIV infection.
* Evidence of viral, bacterial, or fungal infection in the planned treatment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain Measured by the Numerical Rating Scale (NRS) | Days -5 to -1 predosing and days 3 to 14 postdosing
  • Change from baseline of the average daily NRS pain score (scale of 0 to 10 ) of Placebo compared to Active NP2 cohorts.

SECONDARY OUTCOMES:
Opioid Pain Medication Usage Morphine Equivalent Units (MEU) | Days -5 to -1 predosing and 3 to 14 postdosing
  •Change from baseline of use of opioid pain medication average daily MEU of Placebo compared to Active NP2 cohorts
Quality of Life ECOG | Baseline and Week 1, 2 and 4
  •Quality of Life measured by Eastern Cooperative Oncology Group Performance Status (ECOG) assessment at follow-up visits compared to baseline of Placebo compared to Active NP2 cohorts.
Quality of Life SF-12 | Baseline and Week 1, 2 and 4
  •Quality of Life measured by the 12-Item Short Form Health Survey (SF-12v2) at follow-up visits compared to baseline of Placebo compared to Active NP2 cohorts.
Pain SF-MPQ | Baseline and Week 1, 2 and 4
  •Short Form McGill Pain Questionnaire (SF-MPQ-2) assessment at follow-up visits compared to baseline of Placebo compared to Active NP2 cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wolfe, Ph.D., Study Director — Diamyd Inc; David Fink, M.D., Principal Investigator — University of Michigan
Locations (18):
- United States (18):
  - HOPE Research Institute, Phoenix, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Compassionate Cancer Care Medical Group, Inc., Corona, California
  - Cancer Care Associates, Fresno, California
  - TriWest Research Associates, La Mesa, California
  - White Memorial Medical Center, Los Angeles, California
  - Hematology Oncology Associates, Oakland, California
  - Advanced Pharma CR, Miami, Florida
  - Better Health Clinical Research Inc, Newnan, Georgia
  - Christie Clinic, Champaign, Illinois
  - Global Scientific Innovations, Evansville, Indiana
  - Montana Cancer Institute Foundation, Missoula, Montana
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Signal Point Clinical research Center, Middletown, Ohio
  - Pain Research of Oregon, Eugene, Oregon
  - Hematology Oncology Associatesof Rhode Island, Cranston, Rhode Island
  - Medical Therapy and Research, San Antonio, Texas
  - Medical Oncology Associates, Spokane, Washington